CLINICAL TRIAL: NCT07208123
Title: A Bidirectional Cohort Study of Single-Cell Sequencing and Single-Cell Spatial Transcriptomics in Chronic COPD
Brief Title: Mechanistic Studies of Chronic COPD Using Single-Cell Sequencing and Single-Cell Spatial Transcriptomics
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Fang Chen, professor, Tongji University
Other Study IDs: HSCRNACOPD-001
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- COPD group

SUMMARY:
This study is an ambispective cohort study, the sample from patients were from both previously stored and freshly collected . The objective of this study is to investigate the molecular pathological changes underlying the development of chronic obstructive pulmonary disease (COPD). We will use single cell sequencing technology to analyze lung tissue samples from patients who underwent lung resection, with lung tissue from patients without COPD serving as controls. This research aims to provide insights into the pathogenesis of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Receiving lung resection surgery at the hospital for any reason；
* Diagnosed with COPD according to the 2024 GOLD guidelines；
* Tissue samples that meet collection requirements and are either agreed to be collected or already preserved；

Exclusion Criteria:

* Improper preservation of pathological specimens, refusal to consent to sample collection, or incomplete clinical information；
* Combined with other factors causing obstructive airflow limitation;
* Diagnosed with asthma according to the GINA 2023 guidelines and with a history of asthma exacerbations within the past year;
* Combined with Advanced lung cancer;
* Receiving systemic immunosuppressive medications such as anti-rejection drugs;

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 150
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile analysis of lung tissues | until end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China